CLINICAL TRIAL: NCT00657345
Title: IRS Proteins and Trastuzumab Resistance
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Kathryn Edmiston, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: UM200801
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: trastuzumab; breast cancer; her2 positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: This is a tissue acquisition and collection protocol that will analyze potential cellular changes that occur after treatment with trastuzumab.

SUMMARY:
Significant progress has been made in the treatment of women with Her2 positive breast cancer who are treated with trastuzumab, a humanized monoclonal antibody that inhibits Her2. Despite this progress not all patients with Her2 positive metastatic breast cancer respond to trastuzumab and patients with metastatic disease who do respond usually develop progressive disease during treatment with trastuzumab. The mechanism of such resistance is unknown. We propose to investigate the mechanism of trastuzumab resistance in Her2 positive breast cancer. The hypothesis to be examined in the basic science section of this study is that IRS-1 and IRS-2 are modifiers of HER2 signaling and that these adapter proteins could be predictive indicators of treatment response to Herceptin in patients that are candidates for this targeted therapy. The connection between IRS-1 and IRS-2 expression and Herceptin response and clinical outcome in HER2 positive human breast tumors will be evaluated to determine if IRS expression correlates with resistance to Herceptin therapy and with the aggressive behavior of these tumors. This study will establish if the IRS proteins influence HER2 function in tumors and if they are predictive markers for evaluating treatment options for HER2 positive patients.

DETAILED DESCRIPTION:
Twenty percent of invasive breast cancers overexpress Her2 neu. These breast cancers are more aggressive with a higher relapse rate and shortened overall survival. Trastuzumab is a humanized monoclonal antibody FDA approved for the treatment of Her2 overexpressing breast cancer. Trastuzumab is an active single agent for treating metastatic breast cancer and when combined with chemotherapy improves time to progression and overall survival in women with metastatic her2 overexpressing breast cancer. In the adjuvant setting recent clinical trials have demonstrated improved relapse free survival in patients with high risk node negative and node positive breast cancer. In the neoadjuvant setting in patients with locally advanced breast cancer the response rates are very high with complete pathologic responses in 50-60 % of patients. Although trastuzumab is an essential agent for optimal treatment of Her2 positive breast cancer, not all patients respond and in the metastatic setting trastuzumab is not curative indicating that resistance develops. The mechanism of such resistance is unknown.

The fact that not all HER2-expressing breast cancer tumors respond to Herceptin treatment, and most tumors eventually develop resistance to this drug, underscores the need for additional research into how HER2 functions to promote aggressive behavior in tumors and why some tumors become resistant to Herceptin. Recent reports have implicated the IGF-1 signaling pathway in both the mechanism of HER2 action and in resistance to Herceptin. The IRS proteins are the major downstream effectors of the IGF-1 receptor and they play a critical role in determining the cellular response to IGF-1 stimulation. Therefore, the IRS proteins may also be signaling modifiers of the HER2 receptor and may contribute to Herceptin resistance that results from compensatory signaling through the IGF-1R.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18-70 with breast cancer who have signed an IRB approved consent form.
2. Biopsy proven breast cancer with her 2 overexpression by fluorescence in situ hybridization (FISH).
3. Newly diagnosed patients with Stages 1,2 and 3 breast cancer who will be receiving neoadjuvant chemotherapy prior to breast surgery
4. Normal Left ventricular ejection fraction, as measured by echocardiogram or MUGA scan
5. Normal bone marrow, kidney and liver function
6. No evidence of distant metastatic disease

Exclusion Criteria:

1. Patients with significant cardiac disease including abnormal LVEF, symptomatic coronary artery disease, uncontrolled hypertension.
2. Prior treatment with chemotherapy.
3. Any cancer other than previously treated skin cancer.
4. Breast cancer in a previously irradiated breast.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women age 18-70 with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
A tissue acquisition and collection protocol that will analyze potential cellular changes that occur after treatment with trastuzumab to try to elucidate the mechanism of trastuzumab resistance in patients with HER2-positive breast cancer. | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Edmiston, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Mass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Mohsin SK, Weiss HL, Gutierrez MC, Chamness GC, Schiff R, Digiovanna MP, Wang CX, Hilsenbeck SG, Osborne CK, Allred DC, Elledge R, Chang JC. Neoadjuvant trastuzumab induces apoptosis in primary breast cancers. J Clin Oncol. 2005 Apr 10;23(11):2460-8. doi: 10.1200/JCO.2005.00.661. Epub 2005 Feb 14. PMID 15710948
- [Background] Hurley J, Doliny P, Reis I, Silva O, Gomez-Fernandez C, Velez P, Pauletti G, Powell JE, Pegram MD, Slamon DJ. Docetaxel, cisplatin, and trastuzumab as primary systemic therapy for human epidermal growth factor receptor 2-positive locally advanced breast cancer. J Clin Oncol. 2006 Apr 20;24(12):1831-8. doi: 10.1200/JCO.2005.02.8886. Epub 2006 Mar 20. PMID 16549824
- [Background] Coudert BP, Largillier R, Arnould L, Chollet P, Campone M, Coeffic D, Priou F, Gligorov J, Martin X, Trillet-Lenoir V, Weber B, Bleuse JP, Vasseur B, Serin D, Namer M. Multicenter phase II trial of neoadjuvant therapy with trastuzumab, docetaxel, and carboplatin for human epidermal growth factor receptor-2-overexpressing stage II or III breast cancer: results of the GETN(A)-1 trial. J Clin Oncol. 2007 Jul 1;25(19):2678-84. doi: 10.1200/JCO.2006.09.9994. Epub 2007 May 21. PMID 17515572